CLINICAL TRIAL: NCT03075293
Title: Pain Management of Children With Appendicitis in the Emergency Department (ER)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYMC-82-15
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with appendicitis: All children who came to the ER with appendicitis
  Interventions: Other: Determination of pain management

INTERVENTIONS:
Other: Determination of pain management — Determine of pain management given to children with appendicitis in ER according to their medical records

SUMMARY:
The aim of this retrospective study is to determine the percentage of children with appendicitis who were given analgesics or opioids in the ER, to reduce their pain.

ELIGIBILITY:
Inclusion Criteria:

* Children with appendicitis

Exclusion Criteria:

-

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children with appendicitis admitted to the ER
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-03-26 (Estimated); Primary Completion 2017-07-01 (Estimated); Study Completion 2018-04-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of children given pain medication | One year
  Percentage of children given pain medication will be determined according to the data found in their medical records

CONTACTS AND LOCATIONS:
Overall Officials: Muna Kanaani, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No